CLINICAL TRIAL: NCT01951950
Title: Nicardipine Versus Esmolol for Management of Emergence Hypertension After Craniotomy
Brief Title: Nicardipine vs Esmolol Craniotomy Emergence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, John Bebawy, Assistant Professor of Anesthesiology & Neurological Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00083793
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Brain Tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Nicardipine; esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicardipine (Active Comparator): Subjects will receive a 15 mcg/kg bolus of nicardipine as needed followed by an infusion initiated at 5 mg/hr. Nicardipine may be titrated every 5 minutes, increasing 5 mg/hr and administering 15 mcg/kg bolus every minute to a maximum dose of 15 mg/hr. If systolic blood pressure (SBP) is not maintained < 140 mmHg 5 minutes after achieving the maximum dose of nicardipine, medication "failure" will be declared and rescue drug (medication to be determined per anesthesiologist discretion) will be administered. Infusions may be titrated down if SBP decreases below 90 mmHg.
  Interventions: Drug: Nicardipine
- Esmolol (Active Comparator): Subjects will receive a 0.5 mg/kg bolus of esmolol as needed followed by an infusion initiated at 50 mcg/kg/min. Esmolol may be titrated every 5 minutes, increasing 50 mcg/kg/min and administering 0.5 mg/kg bolus every minute to a maximum dose of 200 mcg/kg/min. If SBP is not maintained < 140 mmHg 5 minutes after achieving the maximum dose of esmolol, medication "failure" will be declared and rescue drug (medication to be determined per anesthesiologist discretion) will be administered. Infusions may be titrated down if SBP decreases below 90 mmHg.
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Nicardipine
  Arms: Nicardipine
Drug: Esmolol
  Arms: Esmolol

SUMMARY:
Emergence hypertension is a common occurrence in patients emerging from general anesthesia. This elevation of arterial pressure is particularly concerning in patients undergoing craniotomy due to increased risk of morbidity and mortality in patients with altered intracranial elastance. Thus, identifying better methods to attenuate the hemodynamic changes associated with emergence from anesthesia can improve patient safety, especially in the neurosurgical patient.

Study Hypothesis: Nicardipine is more effective than esmolol as a sole agent in maintaining blood pressure within goal range in the setting of emergence hypertension after craniotomy.

DETAILED DESCRIPTION:
Emergence hypertension following craniotomy is a well-described, albeit poorly understood, phenomenon. Strict control of blood pressure is of utmost importance during and after neurosurgical procedures; failure to prevent acute rises in arterial blood pressure places patients at increased risk of intracranial bleeding, cerebral edema, increased intracranial pressure, and prolonged hospital stays. Emergence hypertension after craniotomy seems to be the result of an acute and transient increase in catecholamine release, peripheral vasoconstriction, and reduced baroreceptor sensitivity. Prior investigations have demonstrated that treatment with antihypertensive agents is required in 60 to 90% of neurosurgical patients postoperatively. Given the common occurrence of emergence hypertension after craniotomy and the increased risk of potentially devastating events that may occur in the setting of acute increases in arterial blood pressure, it is important to identify how best to manage these hemodynamic changes.

An ideal drug for the management of emergence hypertension would be a short-acting, parenteral drug that is easily and rapidly titratable. Medications commonly utilized include nicardipine, labetolol, and esmolol. When given as a bolus, nicardipine, a calcium channel blocker, demonstrates a maximal response in <2 minutes and a mean half-life of approximately 40 minutes. Nicardipine is also frequently administered as an infusion; however, time to onset is increased if no bolus is administered and duration of action may be 4-6 hours after prolonged infusion. Labetolol, a non-selective beta-blocker, demonstrates onset in 10-20 seconds with peak activity at 5 minutes. Esmolol is an ultra-short-acting, B1-beta-blocker that has rapid onset and is quickly metabolized by nonspecific red blood cell esterases; however, esmolol primarily results in decreased heart rate and demonstrates less effect on blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* non-pregnant patients
* (age ≥ 18 years)
* undergoing general anesthesia for elective supratentorial, infratentorial, or transsphenoidal craniotomy

Exclusion Criteria:

* Patients under 18 years of age
* non-English speaking, pregnancy
* emergent craniotomy (including trauma)
* awake craniotomy
* active 3 vessel coronary artery disease or left main coronary artery disease
* advanced heart block
* severe aortic stenosis
* chronic renal failure
* known or suspected allergy or intolerance to a study drug or its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Bebawy, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Bekker A, Didehvar S, Kim S, Golfinos JG, Parker E, Sapson A, Haile M, Kline R, Lee M. Efficacy of clevidipine in controlling perioperative hypertension in neurosurgical patients: initial single-center experience. J Neurosurg Anesthesiol. 2010 Oct;22(4):330-5. doi: 10.1097/ANA.0b013e3181e3077b. PMID 20622687
- [Background] Aronson S, Dyke CM, Stierer KA, Levy JH, Cheung AT, Lumb PD, Kereiakes DJ, Newman MF. The ECLIPSE trials: comparative studies of clevidipine to nitroglycerin, sodium nitroprusside, and nicardipine for acute hypertension treatment in cardiac surgery patients. Anesth Analg. 2008 Oct;107(4):1110-21. doi: 10.1213/ane.0b013e31818240db. PMID 18806012
- [Background] Kross RA, Ferri E, Leung D, Pratila M, Broad C, Veronesi M, Melendez JA. A comparative study between a calcium channel blocker (Nicardipine) and a combined alpha-beta-blocker (Labetalol) for the control of emergence hypertension during craniotomy for tumor surgery. Anesth Analg. 2000 Oct;91(4):904-9. doi: 10.1097/00000539-200010000-00024. PMID 11004045
- [Background] Bilotta F, Lam AM, Doronzio A, Cuzzone V, Delfini R, Rosa G. Esmolol blunts postoperative hemodynamic changes after propofol-remifentanil total intravenous fast-track neuroanesthesia for intracranial surgery. J Clin Anesth. 2008 Sep;20(6):426-30. doi: 10.1016/j.jclinane.2008.04.006. PMID 18929282
- [Background] Kovac AL, Masiongale A. Comparison of nicardipine versus esmolol in attenuating the hemodynamic responses to anesthesia emergence and extubation. J Cardiothorac Vasc Anesth. 2007 Feb;21(1):45-50. doi: 10.1053/j.jvca.2006.08.005. Epub 2006 Oct 24. PMID 17289479

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicardipine: Subjects will receive a 15 mcg/kg bolus of nicardipine as needed followed by an infusion initiated at 5 mg/hr. Nicardipine may be titrated every 5 minutes, increasing 5 mg/hr and administering 15 mcg/kg bolus every minute to a maximum dose of 15 mg/hr. If SBP is not maintained < 140 mmHg 5 minutes after achieving the maximum dose of nicardipine, medication "failure" will be declared and rescue drug (medication to be determined per anesthesiologist discretion) will be administered. Infusions may be titrated down if SBP decreases below 90 mmHg.
Period: Overall Study
Arm/Group | Nicardipine | Esmolol
Started | 26 | 26
Completed | 20 | 20
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicardipine | Esmolol | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (12.7) | 55.9 (12.6) | 56.4 (12.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Failure of Drug to Control Systolic Blood Pressure (SBP) < 140 mmHg
Time Frame: 1 hour postoperatively
Measure: Number; unit: participants
Arm/Group | Nicardipine | Esmolol
Number analyzed (Participants) | 20 | 20
participants | 1 | 11

ADVERSE EVENTS:
Arm/Group | Nicardipine | Esmolol
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes